CLINICAL TRIAL: NCT05598346
Title: Significance and Biological Importance of Mucosal Associated Invariant T Cells in Inflammatory Bowel Disease Patients
Brief Title: Significance of MAIT Cells in Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AL shimaa Mohamed salahidden, principle investigator, Assiut University
Other Study IDs: MAIT cells in In IBD
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Mucosal Associated Invariant T Cells
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To examine the level and function of MAIT cells in IBD patients, and to compare it with disease activity.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBDs), including ulcerative colitis (UC) and Crohn's disease (CD), are chronic inflammatory diseases of unknown origin. IBD has become a global disease with increasing incidence in newly industrialized and westernized countries. Genetic and environmental factors with inadequate host immune response to gut flora appear to play important roles in the pathogenesis of IBD. Adaptive immune response has been classically considered to play a major role in IBD pathogenesis .

Infiltrating lymphocytes including T helper (Th) 1 cells and Th17 cells can lead to the development of intestinal lesions . However, recent evidences suggest that innate immune response is equally important in inducing gut inflammation . Altered epithelial barrier function and aberrant innate immune responses contribute to intestinal inflammation in IBD patients.

Mucosal-associated invariant T (MAIT) cells are innate lymphocytes that express a conserved invariant Tcell receptor (TCR) Vα7.2-Jα33 chain paired with a limited set of Vβ chains. Using distinct pairs of TCR chains, MAIT cells can recognize bacteria-derived riboflavin (vitamin B2) metabolites presented by MHC(major histocompatibility complex) class 1b-like related protein (MR1).

Upon MR1-dependent recognition of antigens, MAIT cells are activated to rapidly release Th1/Th17 proinflammatory cytokines (i.e., interferon [IFN]-γ, tumor necrosis factor [TNF]-α, and interleukin [IL]-17 and cytotoxic molecules (i.e.,granzyme and perforin) to kill infected host cells.

MAIT cells are abundant in peripheral blood where they where they express gut-homing chemokine receptors such as CCR6(chemokine receptor type 6) and CCR9(chemokine receptor type9). They are also abundant in intestinal mucosa where they likely confront normal flora or pathogenic bacteria producing bacterial ligands.

Given tissue- homing properties and rapid production of proinflammatory cytokines, MAIT cells may play an important role in infectious diseases and autoimmune disorders.

Results from experiment with transfer of MAIT cells to TNBS(trinitrobenzene sulfonic acid)-induced IBD murine models suggest that MAIT cells might play a protective role in TNBS-induced intestinal inflammation . In addition, previous studies have reported MAIT cell dysfunction in IBD patients. However, the role of MAIT cells in IBD patients remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active IBD according to clinical scores with the following:

  1. Recently discovered.
  2. Average age (15-50).

Exclusion Criteria:

* Patient with history of any of the following ;

  1. History of respiratory disorders such as chronic obstructive diseases, pulmonary disease or pulmonary embolism.
  2. Other Autoimmune diseases, infectious diseases.
  3. Recent surgery, malignancies, left ventricular dysfunction, use of immunosuppressive drugs.
  4. Chronic liver, renal, and endocrine diseases.

Ages: 15 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Group of patients with active IBD according to clinical scores aged (15-50) , Another group of healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Detection of MAIT cells level in IBD,Compare its level with disease activity | Baseline
  Monoclonal Antibodies by flow cytometry used for detection of MAIT cells in IBD patients

REFERENCES:
- [Result] Xavier RJ, Podolsky DK. Unravelling the pathogenesis of inflammatory bowel disease. Nature. 2007 Jul 26;448(7152):427-34. doi: 10.1038/nature06005. PMID 17653185
- [Result] Garrett WS, Gordon JI, Glimcher LH. Homeostasis and inflammation in the intestine. Cell. 2010 Mar 19;140(6):859-70. doi: 10.1016/j.cell.2010.01.023. PMID 20303876
- [Result] Fonseca-Camarillo G, Yamamoto-Furusho JK. Immunoregulatory Pathways Involved in Inflammatory Bowel Disease. Inflamm Bowel Dis. 2015 Sep;21(9):2188-93. doi: 10.1097/MIB.0000000000000477. PMID 26111210
- [Result] Zhang YZ, Li YY. Inflammatory bowel disease: pathogenesis. World J Gastroenterol. 2014 Jan 7;20(1):91-9. doi: 10.3748/wjg.v20.i1.91. PMID 24415861
- [Result] Giuffrida P, Corazza GR, Di Sabatino A. Old and New Lymphocyte Players in Inflammatory Bowel Disease. Dig Dis Sci. 2018 Feb;63(2):277-288. doi: 10.1007/s10620-017-4892-4. Epub 2017 Dec 23. PMID 29275447
- [Result] Geremia A, Biancheri P, Allan P, Corazza GR, Di Sabatino A. Innate and adaptive immunity in inflammatory bowel disease. Autoimmun Rev. 2014 Jan;13(1):3-10. doi: 10.1016/j.autrev.2013.06.004. Epub 2013 Jun 15. PMID 23774107
- [Result] Treiner E, Duban L, Bahram S, Radosavljevic M, Wanner V, Tilloy F, Affaticati P, Gilfillan S, Lantz O. Selection of evolutionarily conserved mucosal-associated invariant T cells by MR1. Nature. 2003 Mar 13;422(6928):164-9. doi: 10.1038/nature01433. PMID 12634786
- [Result] Kjer-Nielsen L, Patel O, Corbett AJ, Le Nours J, Meehan B, Liu L, Bhati M, Chen Z, Kostenko L, Reantragoon R, Williamson NA, Purcell AW, Dudek NL, McConville MJ, O'Hair RA, Khairallah GN, Godfrey DI, Fairlie DP, Rossjohn J, McCluskey J. MR1 presents microbial vitamin B metabolites to MAIT cells. Nature. 2012 Nov 29;491(7426):717-23. doi: 10.1038/nature11605. Epub 2012 Oct 10. PMID 23051753
- [Result] Napier RJ, Adams EJ, Gold MC, Lewinsohn DM. The Role of Mucosal Associated Invariant T Cells in Antimicrobial Immunity. Front Immunol. 2015 Jul 6;6:344. doi: 10.3389/fimmu.2015.00344. eCollection 2015. PMID 26217338
- [Result] Le Bourhis L, Martin E, Peguillet I, Guihot A, Froux N, Core M, Levy E, Dusseaux M, Meyssonnier V, Premel V, Ngo C, Riteau B, Duban L, Robert D, Huang S, Rottman M, Soudais C, Lantz O. Antimicrobial activity of mucosal-associated invariant T cells. Nat Immunol. 2010 Aug;11(8):701-8. doi: 10.1038/ni.1890. Epub 2010 Jun 27. PMID 20581831
- [Result] Dusseaux M, Martin E, Serriari N, Peguillet I, Premel V, Louis D, Milder M, Le Bourhis L, Soudais C, Treiner E, Lantz O. Human MAIT cells are xenobiotic-resistant, tissue-targeted, CD161hi IL-17-secreting T cells. Blood. 2011 Jan 27;117(4):1250-9. doi: 10.1182/blood-2010-08-303339. Epub 2010 Nov 17. PMID 21084709
- [Result] Cosgrove C, Ussher JE, Rauch A, Gartner K, Kurioka A, Huhn MH, Adelmann K, Kang YH, Fergusson JR, Simmonds P, Goulder P, Hansen TH, Fox J, Gunthard HF, Khanna N, Powrie F, Steel A, Gazzard B, Phillips RE, Frater J, Uhlig H, Klenerman P. Early and nonreversible decrease of CD161++ /MAIT cells in HIV infection. Blood. 2013 Feb 7;121(6):951-61. doi: 10.1182/blood-2012-06-436436. Epub 2012 Dec 18. PMID 23255555
- [Result] Leeansyah E, Ganesh A, Quigley MF, Sonnerborg A, Andersson J, Hunt PW, Somsouk M, Deeks SG, Martin JN, Moll M, Shacklett BL, Sandberg JK. Activation, exhaustion, and persistent decline of the antimicrobial MR1-restricted MAIT-cell population in chronic HIV-1 infection. Blood. 2013 Feb 14;121(7):1124-35. doi: 10.1182/blood-2012-07-445429. Epub 2012 Dec 13. PMID 23243281
- [Result] Meierovics AI, Cowley SC. MAIT cells promote inflammatory monocyte differentiation into dendritic cells during pulmonary intracellular infection. J Exp Med. 2016 Nov 14;213(12):2793-2809. doi: 10.1084/jem.20160637. Epub 2016 Oct 31. PMID 27799620
- [Result] Meierovics A, Yankelevich WJ, Cowley SC. MAIT cells are critical for optimal mucosal immune responses during in vivo pulmonary bacterial infection. Proc Natl Acad Sci U S A. 2013 Aug 13;110(33):E3119-28. doi: 10.1073/pnas.1302799110. Epub 2013 Jul 29. PMID 23898209
- [Result] Grimaldi D, Le Bourhis L, Sauneuf B, Dechartres A, Rousseau C, Ouaaz F, Milder M, Louis D, Chiche JD, Mira JP, Lantz O, Pene F. Specific MAIT cell behaviour among innate-like T lymphocytes in critically ill patients with severe infections. Intensive Care Med. 2014 Feb;40(2):192-201. doi: 10.1007/s00134-013-3163-x. Epub 2013 Dec 10. PMID 24322275
- [Result] Jiang J, Wang X, An H, Yang B, Cao Z, Liu Y, Su J, Zhai F, Wang R, Zhang G, Cheng X. Mucosal-associated invariant T-cell function is modulated by programmed death-1 signaling in patients with active tuberculosis. Am J Respir Crit Care Med. 2014 Aug 1;190(3):329-39. doi: 10.1164/rccm.201401-0106OC. PMID 24977786
- [Result] Kim JC, Jin HM, Cho YN, Kwon YS, Kee SJ, Park YW. Deficiencies of Circulating Mucosal-associated Invariant T Cells and Natural Killer T Cells in Patients with Acute Cholecystitis. J Korean Med Sci. 2015 May;30(5):606-11. doi: 10.3346/jkms.2015.30.5.606. Epub 2015 Apr 15. PMID 25931792
- [Result] Kwon YS, Cho YN, Kim MJ, Jin HM, Jung HJ, Kang JH, Park KJ, Kim TJ, Kee HJ, Kim N, Kee SJ, Park YW. Mucosal-associated invariant T cells are numerically and functionally deficient in patients with mycobacterial infection and reflect disease activity. Tuberculosis (Edinb). 2015 May;95(3):267-74. doi: 10.1016/j.tube.2015.03.004. Epub 2015 Mar 21. PMID 25837440
- [Result] Miyazaki Y, Miyake S, Chiba A, Lantz O, Yamamura T. Mucosal-associated invariant T cells regulate Th1 response in multiple sclerosis. Int Immunol. 2011 Sep;23(9):529-35. doi: 10.1093/intimm/dxr047. Epub 2011 Jun 28. PMID 21712423
- [Result] Cho YN, Kee SJ, Kim TJ, Jin HM, Kim MJ, Jung HJ, Park KJ, Lee SJ, Lee SS, Kwon YS, Kee HJ, Kim N, Park YW. Mucosal-associated invariant T cell deficiency in systemic lupus erythematosus. J Immunol. 2014 Oct 15;193(8):3891-901. doi: 10.4049/jimmunol.1302701. Epub 2014 Sep 15. PMID 25225673
- [Result] Serriari NE, Eoche M, Lamotte L, Lion J, Fumery M, Marcelo P, Chatelain D, Barre A, Nguyen-Khac E, Lantz O, Dupas JL, Treiner E. Innate mucosal-associated invariant T (MAIT) cells are activated in inflammatory bowel diseases. Clin Exp Immunol. 2014 May;176(2):266-74. doi: 10.1111/cei.12277. PMID 24450998
- [Result] Ruijing X, Mengjun W, Xiaoling Z, Shu P, Mei W, Yingcheng Z, Yuling H, Jinquan T. Jalpha33+ MAIT cells play a protective role in TNBS induced intestinal inflammation. Hepatogastroenterology. 2012 May;59(115):762-7. doi: 10.5754/hge11432. PMID 22115767
- [Result] Walsh AJ, Ghosh A, Brain AO, Buchel O, Burger D, Thomas S, White L, Collins GS, Keshav S, Travis SP. Comparing disease activity indices in ulcerative colitis. J Crohns Colitis. 2014 Apr;8(4):318-25. doi: 10.1016/j.crohns.2013.09.010. Epub 2013 Oct 10. PMID 24120021
- [Result] Feagan BG, Sandborn WJ, D'Haens G, Panes J, Kaser A, Ferrante M, Louis E, Franchimont D, Dewit O, Seidler U, Kim KJ, Neurath MF, Schreiber S, Scholl P, Pamulapati C, Lalovic B, Visvanathan S, Padula SJ, Herichova I, Soaita A, Hall DB, Bocher WO. Induction therapy with the selective interleukin-23 inhibitor risankizumab in patients with moderate-to-severe Crohn's disease: a randomised, double-blind, placebo-controlled phase 2 study. Lancet. 2017 Apr 29;389(10080):1699-1709. doi: 10.1016/S0140-6736(17)30570-6. Epub 2017 Apr 12. PMID 28411872
- [Result] Gajendran M, Loganathan P, Catinella AP, Hashash JG. A comprehensive review and update on Crohn's disease. Dis Mon. 2018 Feb;64(2):20-57. doi: 10.1016/j.disamonth.2017.07.001. Epub 2017 Aug 18. PMID 28826742